CLINICAL TRIAL: NCT03903393
Title: Serum LncRNAs as Early Potential Biomarkers for the Prediction of Preeclampsia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 201933
Record Dates: First submitted 2019-04-03; First posted 2019-04-04 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-03

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. the serum of the pregnant women
  2. the placenta of the pregnant women after delivery
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- preeclamptic women: systolic blood pressure(BP) ≥140 mm Hg or diastolic BP ≥90 mm Hg; hypertension diagnosed after 20 weeks gestation; new-onset hypertension with new-onset proteinuria or other signs/symptoms of preeclampsia after 20 weeks or chronic proteinuria with newonset hypertension.
- controls: Normal pregnant women

SUMMARY:
To identify lncRNAs differentially expressed at early stages of gestation in the serum of pregnant women, who later developed severe preeclampsia (sPE) in the third trimester of pregnancy compared to women with normal pregnancy .

DETAILED DESCRIPTION:
Preeclampsia (PE) is a pregnancy syndrome characterized by hypertension and proteinuria, and a leading cause of maternal and fetal morbidity and mortality, with poorly defined pathophysiological mechanisms remain. Circulating lncRNAs are long, noncoding RNA molecules, which negatively regulate gene expression, and considered as promising biomarkers for PE. The objective of the study is to evaluate circulating lncRNA signatures in women with PE compared to healthy women, and in women sub-grouped per PE severity. This study assessed lncRNA expression profile in the serum at early stages of gestation of women who later developed severe preeclampsia (sPE) in the third trimester of pregnancy compared to women with uncomplicated pregnancies. Circulating lncRNA was extracted from maternal serum. This study also assess lncRNA expression profile in the placenta tissues of PE patients and healthy pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* new onset hypertension (systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg on two occasions at least 4 h apart) after 20 weeks of gestation in women who previously had normal blood pressure.
* proteinuria (the excretion of 300 mg or more of protein in a 24-hour urine collection)or other signs/symptoms of preeclampsia after 20 weeks of gestation in women who previously had normal blood pressure.

Exclusion Criteria:

* maternal infections
* smoking
* chemical dependency
* known major foetal or chromosomal anomalies
* intrahepatic cholestasis during pregnancy
* assisted reproductive technology (ART) treatments
* chronic hypertension.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Preeclamptic women Controls
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2019-03-31 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
The RNA expression levels of lncRNAs | 5 months
  the serum of patients with preeclampsia and in the serum of normal controls were measured by qRT-PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Yue Li, Principal Investigator — First Affiliated Hospital of Harbin Medical University
Locations (1):
- Serum LncRNAs as Potential Biomarkers for the Prediction of Preeclampsia, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Undecided